CLINICAL TRIAL: NCT04857853
Title: Effects of Exercise, Rest Breaks and Ergonomics Modification on Fatigue and Musculoskeletal Discomfort in Static Workstation Office Workers
Brief Title: Exercise, Rest Breaks and Ergonomics Modification on Fatigue and MSK Discomfort in Static Workstation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00858 Anam Rehman
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Musculoskeletal Pain
Keywords: Pain; Workstation; Musculoskeletal; Rest break
MeSH Terms: conditions — Musculoskeletal Pain; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Without Rest Breaks (Experimental): Exercise Without Rest Breaks
  Interventions: Other: Exercise Without Rest Break
- Exercise With Rest Break (Experimental): Exercise With Rest Break
  Interventions: Other: Exercise With Rest Break
- Rest Break (Experimental): Rest Break
  Interventions: Other: Rest Break

INTERVENTIONS:
Other: Exercise Without Rest Break — Participants in the exercise group will receive 'Exercise Breaks', of 10 minutes, twice a day during the work hours, in addition to the two 'Conventional Rest Breaks' of 15 minutes, twice a day during the work hours.
  Exercises include shoulder shrugs, neck tilts, wrist and forearm stretch, back and hip stretch, upper body stretch, hamstring stretch, upper back stretch, hand/finger stretch. Side stretch and neck stretch.
  Follow up 3 times a week for 5 weeks.
  Arms: Exercise Without Rest Breaks
Other: Exercise With Rest Break — Participants in the exercise with rest break group will receive 'Exercise Breaks', of 10 minutes, twice a day during the work hours, in addition to the two 'Conventional Rest Breaks' of 15 minutes, twice a day during the work hours.
  Participants will also receive 'Supplemental Micro Breaks', of 30 seconds after every 15 minutes of working on a static computer workstation Follow up 3 times a week for 5 weeks.
  Arms: Exercise With Rest Break
Other: Rest Break — Participants in the rest breaks group will receive 'Supplemental Micro Breaks', of 30 seconds after every 15 minutes of working on a static computer workstation in addition to the two 'Conventional Rest Breaks' of 15 minutes twice a day during the work hours.
  Follow up 3 times a week for 5 weeks. During the rest breaks, participants will not perform any exercises.
  Arms: Rest Break

SUMMARY:
The current study examines the effects of exercise, ergonomic modifications, and rest breaks on fatigue and musculoskeletal discomfort during computer tasks. For the purpose of this project, musculoskeletal discomfort is defined as a constellation of signs and symptoms that include muscle tension, paresthesia, pain, and/or physical strain in soft tissues and bones.

DETAILED DESCRIPTION:
Static workstation workers frequently experience musculoskeletal discomfort which, according to a survey of the literature, may include muscle tension, muscle fatigue, paresthesia, pain, and/or physical strain in soft tissues and bones. The incidence of musculoskeletal discomfort in office workers like computer users is as high as 50%. In various studies on static workstation workers, musculoskeletal discomfort has been reported, either separately or in aggregate, in the neck, shoulders, elbows, wrists, hands, back, legs, buttocks, ankles, feet, and chest.

The current study examines the effects of exercise, ergonomic modifications, and rest breaks on fatigue and musculoskeletal discomfort during computer tasks. For the purpose of this project, musculoskeletal discomfort is defined as a constellation of signs and symptoms that include muscle tension, paresthesia, pain, and/or physical strain in soft tissues and bones.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age: 25-45 years
* Those static workstation office workers using a computer for at least 6 hours per day.
* Static workstation office workers screened by ROSA.

Exclusion Criteria:

* Discomfort from non-musculoskeletal origin
* Recent history of trauma and receiving any kind of treatment for the current condition
* Severe orthopedic disease
* Any mental and physiological illness that could interfere in the exercise

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal Discomfort Questionnaire | 6th week
  To assess the severity of musculoskeletal discomfort. minimum as Never = 0, and maximum as Several times every day = 10 The discomfort score is the severity of discomfort categorized as 'mild', 'moderate', and 'severe discomfort'.
Chalder fatigue scale | 6th week
  Each of the 11 items is answered on a 4-point scale ranging from the asymptomatic to maximum symptomology, such as 'Better than usual', 'No worse than usual, 'Worse than usual, and 'Much worse than usual.

CONTACTS AND LOCATIONS:
Overall Officials: Nazish Rafique, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Foundation University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarwaka P, Bakri LS. Ergonomi Industri Dasar-dasar pengetahuan ergonomi dan aplikasi di tempat kerja. Surakarta: Harapan Press; 2010.
- [Background] Daneshmandi H, Choobineh AR, Ghaem H, Alhamd M, Fakherpour A. The effect of musculoskeletal problems on fatigue and productivity of office personnel: a cross-sectional study. J Prev Med Hyg. 2017 Sep;58(3):E252-E258. PMID 29123372
- [Background] Rahimi R. Effect of different rest intervals on the exercise volume completed during squat bouts. J Sports Sci Med. 2005 Dec 1;4(4):361-6. eCollection 2005 Dec. PMID 24501549
- [Background] Barredo RDV, Mahon K. The effects of exercise and rest breaks on musculoskeletal discomfort during computer tasks: An evidence-based perspective. Journal of Physical Therapy Science. 2007;19(2):151-63.
- [Background] Willardson JM, Burkett LN. A comparison of 3 different rest intervals on the exercise volume completed during a workout. J Strength Cond Res. 2005 Feb;19(1):23-6. doi: 10.1519/R-13853.1. PMID 15705039
- [Background] Menzel NN, Brooks SM, Bernard TE, Nelson A. The physical workload of nursing personnel: association with musculoskeletal discomfort. Int J Nurs Stud. 2004 Nov;41(8):859-67. doi: 10.1016/j.ijnurstu.2004.03.012. PMID 15476759
- [Background] Hamberg-van Reenen HH, van der Beek AJ, Blatter BM, van der Grinten MP, van Mechelen W, Bongers PM. Does musculoskeletal discomfort at work predict future musculoskeletal pain? Ergonomics. 2008 May;51(5):637-48. doi: 10.1080/00140130701743433. PMID 18432442
- [Background] Hou JY, Shiao JS. Risk factors for musculoskeletal discomfort in nurses. J Nurs Res. 2006 Sep;14(3):228-36. doi: 10.1097/01.jnr.0000387581.04716.56. PMID 16967405